CLINICAL TRIAL: NCT05324527
Title: The Effect of Preoperational Hand Massage Applied to Children on Anxiety Level And Hemodynamic Variables: A Randomized Controlled Trial
Brief Title: The Effect of Preoperational Hand Massage Anxiety Level And Hemodynamic Variables
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Didem Lafci, PhD, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MersinUniv
Record Dates: First submitted 2022-03-25; First posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Anxiety; Hemodynamic Instability
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, two-arm, randomized controlled clinical trial
Who Masked: Participant
Masking Description: Masking Description According to the randomization table, the information showing the patients included in the research sample is assigned to the A and B groups will be put in an opaque envelope. This envelope will be kept by the coordinator researcher (DL) and when the researcher (FA) goes to the patient for application, after filling out the "Informed Voluntary Consent Form", he will open the envelope and learn which group is in which group. Due to the nature of the study, patients and the researcher (FA) will notbe blinded, since abdominal massage will be applied only to the patients included in the study. When the research is completed, the data will be transferred to the computer environment by a statistician who does not know the A and B groups, and the data will be analyzed by a statistician independent of the research and the findings will be reported. Thus, the data analysis and statistics phase will be blind to group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand Massage Group (Experimental): After the researcher and the children in study group sat on a chair facing each other, hand massage procedure, 8 minutes to both hands and a total of 16 minutes hand massage was applied with liquid petrolatum.
  Interventions: Other: Hand Massage
- Control group (No Intervention): The control group will be received routine treatment and care in the unit.

INTERVENTIONS:
Other: Hand Massage — Hand massage procedure, 8 minutes to both hands and a total of 16 minutes hand massage was applied with liquid petrolatum.
  Arms: Hand Massage Group

SUMMARY:
The study was conducted randomly controlled experimental to determine the effect of hand massage applied to pre-operative children on anxiety level and physical symptoms of anxiety.

DETAILED DESCRIPTION:
On operation morning, "Child and Parent Introduction Form", "State-Trait Anxiety Inventory for Children" were read to and "Physiological Symptoms of Anxiety Inspection Form" measurement was done on children in both groups, and their 1st measurement values were recorded. Routine treatment and nursing care applications of the service were done preoperationally. After the researcher and the children in study group sat on a chair facing each other, hand massage procedure, 8 minutes to both hands and a total of 16 minutes hand massage was applied with liquid petrolatum. No massage was applied to children in control group. Right 16 minutes after the 1st filled forms in each group, "State-Trait Anxiety Inventory for Children", "Physiological Symptoms of Anxiety Inspection Form" were read, measurement was done and 2nd measurement values were recorded. Furthermore, "Satisfaction Evaluation Scale" was marked by those in study group after the massage, and measurement values were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the study and obtaining written permission from the family,
* Able to speak and understand Turkish,
* Not taking any analgesic and anesthetic drugs before the procedure,
* Over 9 years old and under 12 years old,
* whose parents are literate,
* Poor general condition and not needing emergency surgery (cases such as acute abdomen, intestinal perforations, traumas, etc.),
* There is no open wound on the skin or an obstacle to massage (edema, abscess, skin infection with necrosis, etc.),
* Thrombophlebitis, occlusive artery disease, fever etc. who do not have a situation in which massage application is objectionable due to illness, He does not have conditions such as loss of sensation, mass, fracture and ingrown nails in his hand,
* Children who are conscious, fully oriented and cooperative and open to communication

Exclusion Criteria:

* Those who do not accept to participate in the research and do not get written permission from their families,
* Does not speak or understand Turkish
* Taking any analgesic and anesthetic drugs before the procedure,
* Less than 9 years old and over 12 years old,
* illiterate parents
* Poor general condition and emergency surgery (acute abdomen, intestinal perforations, traumas, etc.) cases) need,
* Open wound on the skin or an obstacle to massage (edema, abscess, necrosis has occurred) skin infection etc.)
* Thrombophlebitis, occlusive artery disease, fever etc. massage practice due to illness having a situation where it is objectionable,
* Having conditions such as loss of sensation in the hand, mass, fracture and ingrown nails,
* Children who are unconscious, oriented and cooperative and not open to communication

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Anxiety evaluated using the State Anxiety Scale | Change from before implementation and after 16 minutes of practice (hand massage)
  Scores ranging from 20 to 80 points are obtained in the scale. In the total score obtained from the scale in scoring the scale, 0-19 points indicate the absence of anxiety, 20-39 points indicate mild anxiety, 40-59 points indicate moderate anxiety, and 60-79 points indicate severe anxiety level. Higher state anxiety scores indicate that anxiety level is also hig

SECONDARY OUTCOMES:
Blood pressure | Change from before implementation and after 16 minutes of practice (hand massage)
  systolic blood pressure (SBP), diastolic blood pressure (DBP), mmHg
Heart rate | Change from before implementation and after 16 minutes of practice (hand massage)
  beats per minute
respiratory rate | Change from before implementation and after 16 minutes of practice (hand massage)
  ekspiration and inspiration per minute
peripheral oxygen saturation | Change from before implementation and after 16 minutes of practice (hand massage)
  %, percentage of oxygenated hemoglobin in peripheral arterial blood

CONTACTS AND LOCATIONS:
Overall Officials: Fahri AŞKAN, Master, Principal Investigator — 100. Year University
Locations (1):
- Mersin University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No